CLINICAL TRIAL: NCT02702778
Title: A Randomized, Open-label, Dose-ranging Study of Oral Delayed Release Prednisone in Patients With Untreated Polymyalgia Rheumatic (PMR)
Brief Title: Delayed Release Prednisone in PMR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of study recruitment
Sponsor: Dinora, Inc. (Other)
Collaborators: Analgesic Solutions (Industry); PharPoint Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-PRE-IIS02
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica (PMR)
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4mg DR-Prednisone (Active Comparator): Subjects in this arm will receive a night-time dose of 4mg delayed-release prednisone for two weeks followed by treatment with 15mg IR-prednisone in the morning for two weeks.
  Interventions: Drug: Delayed-Release (DR) Prednisone; Drug: Immediate Release (IR) Prednisone
- 7mg DR-Prednisone (Active Comparator): Subjects in this arm will receive a night-time dose of 7mg delayed-release prednisone for two weeks followed by treatment with 15mg IR-prednisone in the morning for two weeks.
  Interventions: Drug: Delayed-Release (DR) Prednisone; Drug: Immediate Release (IR) Prednisone
- 10mg DR-Prednisone (Active Comparator): Subjects in this arm will receive a night-time dose of 10mg delayed-release prednisone for two weeks followed by treatment with 15mg IR-prednisone in the morning for two weeks.
  Interventions: Drug: Delayed-Release (DR) Prednisone; Drug: Immediate Release (IR) Prednisone

INTERVENTIONS:
Drug: Delayed-Release (DR) Prednisone — delayed release prednisone
  Other Names: RAYOS
Drug: Immediate Release (IR) Prednisone — standard prednisone

SUMMARY:
A four-week, randomized, controlled, open-label trial of DR prednisone in which patients receive in period 1 one of three-night time doses of treatment (4mg, 7mg or 10mg) for two weeks followed in period 2 by treatment with 15mg IR prednisone in the morning for two weeks. Period 1 is randomized and open-label and period 2 is open label. Before enrollment and randomization patient diagnosis and responsiveness to 15mg IR prednisone in the morning is established. 45 patients will be randomized, 15 patients in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PMR:

   1. All participants must meet the Bird criteria (7): 3 or more of the following features are required to make the diagnosis.

      * Bilateral shoulder pain/stiffness
      * Onset of symptoms <2 weeks
      * Initial Erythrocyte Sedimentation Rate (ESR) >40 mm/h
      * Stiffness >1 h
      * Age >65 years
      * Depression and/or weight loss
      * Bilateral upper arm tenderness
   2. All participants must have PMR in the opinion of the PI
2. Are over 50 years old.
3. No or stable NSAID or analgesic therapy for at least 7 days.
4. Currently active disease defined by a C-reactive protein (CRP) at least 5mg/L, or ESR at least 29mm in one hour measured at the screening visit or within the previous week.
5. Respond to one week of 15 mg IR prednisone and one week washout (patient worsens). Response will be measured as: >70% reduction in morning stiffness severity at the end of the first week with a >80% return of morning stiffness severity in the second week (screening procedure). This screening procedure can also be assessed in patients who have taken up to one week of >15 mg IR prednisone prior to seeing the investigator for the study, so long as informed consent is obtained before the wash-out period and all other inclusion criteria are met.

Exclusion Criteria:

1. Oral glucocorticoid treatment for more than 1 week within the previous month
2. Parenteral glucocorticoid treatment within the last month
3. Pregnancy and/or lactation
4. Inflammatory diseases such as inflammatory bowel disease, colitis, asthma, rheumatoid arthritis
5. Co-existent giant cell arteritis; patients with headache, visual symptoms or jaw claudication suggestive of giant cell arteritis will not be included in the study
6. Other auto-immune diseases
7. Synovitis or polymyositis
8. Positive Cyclic Citrullinated Peptide Antibodies (CCP)
9. Muscle weak and elevated creatinine phosphokinase (CPK)
10. Cancer (patients with a history of basal cell carcinoma or cancer-free for > 5 years are allowed)
11. Severe active infection including herpes or other viral or bacterial infection(s), treatment with antibiotics within the past 6 weeks or have or had a history of tuberculosis
12. Significant renal disease (creatinine greater than150 µmol/L)
13. Significant hepatic impairment (ALT/AST greater than twice upper limit of normal)
14. Immunization with live vaccines within 8 weeks before the first administration of the study drug or plan to have an immunization with a live vaccine within 2 weeks after the last administration of study drug.
15. Use of any other systemic glucocorticoids including inhalants during the screening and treatment phase of the study; chronic intranasal or ophthalmic corticosteroids are allowed.
16. Participation in a clinical trial of an investigational drug within the past 30 days
17. Working night-time shift employee
18. Jet lag (i.e. airplane travel)
19. Unable to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change of the severity of morning stiffness from baseline to end of study (28days) | Assessed daily from screening through End of Study visit, 28 days total
  To determine the relative reduction in the severity of morning stiffness of three night time doses (4mg, 7mg, and 10mg) of DR prednisone after 2 weeks compared to the reduction after treatment with IR prednisone15mg in the morning for 2 weeks in newly diagnosed PMR patients (with no evidence of other systemic inflammatory diseases such as RA) who are known to be responsive to standard treatment with IR prednisone15mg in the morning. This will be assessed using a 10cm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Relative reduction in the duration of morning stiffness (minutes) | Assessed daily from screening through End of Study visit, an average of 2 months
  This will be assessed via a questionnaire.
Relative IL-6 treatment response. | Assessed at Baseline, Day 14, and Day 28
Changes in plasma IL-6 compared with changes in the severity of morning stiffness | Through study completion, a total of 3 assessments over 28days
Patient reported outcomes in accordance with the OMERACT PMR objectives | Through study completion, an average of 2 months.
Performance characteristics of additional clinical measures of disease outcome. | Through study completion, an average of 2 months
  Additional characteristics such as pain and fatigue will be assessed using a 10cm Visual Analog Scale (VAS).

OTHER OUTCOMES:
Changes in PMR Activity Score (PMRAS) following treatment with DR prednisone and IR prednisone | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Mineola, New York
  - Clinical Research Site, Duncansville, Pennsylvania
  - Clinical Research Site 2, Wyomissing, Pennsylvania
  - Clinical Research Site, Wyomissing, Pennsylvania
  - Clinical Research Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No